CLINICAL TRIAL: NCT05134038
Title: L'impact De La Raideur Articulaire Pelvienne Sur La Peur De Chuter Du Sujet Âgé Hospitalisé Ou En Institution.
Brief Title: Association Between Fear of Falling and Spinal Stiffness.
Acronym: RAAPC
Status: Completed | Type: Observational
Sponsor: Hopital of Melun (Other)
Responsible Party: Principal Investigator, Sebastien Jochmans, MD, Head of Clinical Research Unit, Groupe Hospitalier Sud Ile-de-France
Other Study IDs: 294-URC-GHSIF
Record Dates: First submitted 2021-10-23; First posted 2021-11-24 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Joint(S) Degeneration; Old Age; Atrophy; Fear of Injury
MeSH Terms: conditions — Joint Diseases; Atrophy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: anthropomorphic measurements — anthropomorphic measurements + FES questionnaire + demographic data and medications
  Other Names: FES questionnaire

SUMMARY:
1. / evaluation of the fear of falling using an FES-I questionnaire, distribution of subjects according to the score into 3 groups (16-19: little concerned by the fear of falling, 20-27 moderately concerned, 28-64 very concerned by fear of falling)
2. / evaluation of lumbar articular mobility by the schober index, coxofemoral by hip goniometry in flexion and extension (no evaluation of other amplitudes because lack of abduction / abduction / external and internal rotation of the hip remain functional in walking and the balance)

DETAILED DESCRIPTION:
1. / evaluation of the fear of falling using an FES-I questionnaire, distribution of subjects according to the score into 3 groups (16-19: little concerned by the fear of falling, 20-27 moderately concerned, 28-64 very concerned by fear of falling)
2. / evaluation of lumbar articular mobility by the schober index, coxofemoral by hip goniometry in flexion and extension (no evaluation of other amplitudes because lack of abduction / abduction / external and internal rotation of the hip remain functional in walking and the balance)

ELIGIBILITY:
Inclusion Criteria:

* over 75 years old,
* Ability to understand and answer a questionnaire in French
* Ability to stand up
* Patient from the Melun hospital (santé pole center + nursing home of the GHSIF)
* Affiliated with a social security scheme

Exclusion Criteria:

* mental disorders,
* lumbar surgery

Min Age: 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: > 75 ans, in any geriatric department of the hospital
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Association FES and goniometry | 15 minutes
  Highlight a significant positive association between hips' goniometry (angle degree) and FES-I score (continuous scale without unit)
Association FES-I (continuous scale without unit) and Schober index (centimeter) | 15 minutes
  Highlight a significant positive association between Shober index and FES-I score

CONTACTS AND LOCATIONS:
Overall Officials: SEBASTIEN JOCHMANS, M.D., Study Director — GHSIF MELUN
Locations (1):
- GH Sud Ile-de-France, CH Melun-Sénart, Melun, France, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tinetti ME, Powell L. Fear of falling and low self-efficacy: a case of dependence in elderly persons. J Gerontol. 1993 Sep;48 Spec No:35-8. doi: 10.1093/geronj/48.special_issue.35. No abstract available. PMID 8409238
- [Background] Kendrick D, Kumar A, Carpenter H, Zijlstra GA, Skelton DA, Cook JR, Stevens Z, Belcher CM, Haworth D, Gawler SJ, Gage H, Masud T, Bowling A, Pearl M, Morris RW, Iliffe S, Delbaere K. Exercise for reducing fear of falling in older people living in the community. Cochrane Database Syst Rev. 2014 Nov 28;2014(11):CD009848. doi: 10.1002/14651858.CD009848.pub2. PMID 25432016
- [Background] Delbaere K, Close JC, Mikolaizak AS, Sachdev PS, Brodaty H, Lord SR. The Falls Efficacy Scale International (FES-I). A comprehensive longitudinal validation study. Age Ageing. 2010 Mar;39(2):210-6. doi: 10.1093/ageing/afp225. Epub 2010 Jan 8. PMID 20061508